CLINICAL TRIAL: NCT03557463
Title: Use of UV-treated Milk Powder to Increase Vaccine Efficacy in the Elderly
Brief Title: Testing a Novel Dairy Protein to Counteract Immunosenescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1164896
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Immunodeficiency
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Intervention Model Description: Controlled, randomized, double blind pilot study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Supplements were coded based on protein type and both participants and researchers were blinded to the underlying code
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soy protein (Active Comparator): Low isoflavone soy protein powder: Each participant was required to consume a total of 112 servings for the 8-week duration of the study. A 4-week supply was provided at baseline (week 0) and at the time of vaccine administration (week 4).
  Interventions: Dietary Supplement: Dairy protein
- Dairy protein (Experimental): UV-C treated raw milk protein supplement (TruActiv MPC 85). Each participant was required to consume a total of 112 servings for the 8-week duration of the study. A 4-week supply was provided at baseline (week 0) and at the time of vaccine administration (week 4).
  Interventions: Dietary Supplement: Dairy protein

INTERVENTIONS:
Dietary Supplement: Dairy protein — A controlled, randomized, double blind pilot study was conducted using two different protein sources as nutritional supplementation to enhance vaccine response.

SUMMARY:
Aging populations experience a decline in adaptive immune system function also known as immunosenesence. Nutritional approaches to stimulate and strengthen the immune system are needed for this growing segment of the population. A controlled, randomized, double blind pilot study was conducted using two different protein sources as nutritional supplementation to enhance vaccine response. Our objective was to examine the immune stimulating effects of dairy protein subjected to ultraviolet radiation (UV-C) radiation treatment process instead of pasteurization. Participants were 21 healthy individuals over 60 years of age who consumed 6 g of the dairy protein or a comparison, soy isoflavone protein, twice a day for eight weeks. DTaP vaccine administered at week 4. Non-parametric t-tests revealed a significant increase in Tetanus antibodies in the dairy group compared to the soy group at week 8. These findings suggest additional benefits of UV-C treated unheated dairy protein as a solution to counteract immunosenescence, but warrant further study in elderly and other populations that might benefit from immune system stimulation.

ELIGIBILITY:
Inclusion criteria included participants be more than 60 years of age. Volunteers underwent a physical examination and health assessment by a physician to ensure the absence of exclusion criteria which were regular consumption of greater than one unit of milk and/or milk products (milk, yogurt, fresh cheese, etc.) a day at the time of enrollment, known milk allergy, food faddism, other non-traditional diet, prolonged consumption of dairy supplements (greater than one daily during the previous four weeks), use of tobacco products in the previous 10 years, underlying neoplasia or immunological disease, including hypergammaglobunemia, renal disease or failure, use of steroids or immunosuppressive drugs in the previous eight weeks, reduced physical activity (New York Heart Association classes III-IV). Having received a DTaP vaccine within the last five years was an exclusion criteria for the study, but patient records were incomplete for many volunteers on this aspect. Therefore, volunteers with an initial Tetanus antibody level above 3 IU/mL were excluded from the study results as the volunteer was assumed to have had the DTaP vaccine within the last 5 years.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Immune response to vaccine | 8 weeks
  Difference in DTaP vaccine antibodies at before and after vaccine

IPD SHARING:
Plan to Share IPD: Undecided